CLINICAL TRIAL: NCT01557933
Title: A Study of the Acute and Chronic Effects of Electroconvulsive Therapy on Glutamatergic Neurotransmission in Bipolar Depression
Brief Title: Effects of Electroconvulsive Therapy (ECT) in Bipolar Depression
Status: Withdrawn | Type: Observational
Why Stopped: Due to a lack of participants, this study has been closed.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director for Translational Neuroscience Research, Mclean Hospital
Other Study IDs: 2011-P-000693
Record Dates: First submitted 2012-03-09; First posted 2012-03-20 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Bipolar Disorder
Keywords: ECT; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECT: All study subjects have consented to receive ECT.
  Interventions: Other: No interventions will be used

INTERVENTIONS:
Other: No interventions will be used — No interventions will be used

SUMMARY:
The primary purpose of this study is to use magnetic resonance spectroscopy (MRS) to measure the levels of several brain chemicals including, but not limited to, glutamate, glutamine, and N-acetylaspartate, before and after treatment with ECT. In addition to MRS, the investigators will use several other MRI techniques including structural MRI, resting state functional MRI (fMRI), and diffusion tensor imaging (DTI) to measure how the structure and function of the brain changes with ECT.

The investigators hypothesize that the Gln/Glu ratio is increased in the anterior cingulate cortex (ACC), but not the parieto-occipital cortex (POC), following the first ECT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-55
* Meets DSM-IV criteria for Bipolar Disorder Type I, II, or NOS with current episode depressed
* Has been scheduled to be evaluated by an ECT consultant from the McLean Hospital ECT service
* Current score of greater than or equal to 24 on the Montgomery-Asberg Depression Rating Scale (MADRS)

Exclusion Criteria:

* Unwillingness or inability to provide informed consent
* Lifetime history of schizophrenia
* DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine dependence, within three months prior to screening
* Positive urine toxicology screen at screening (NOTE: Participants with a positive urine toxicology screen who are prescribed benzodiazepine, stimulant, or opiate medications by their physician will be permitted to enroll in the study as long as they do not meet abuse or dependence criteria for these substances)
* Female participants with a positive urine pregnancy test at screening
* Pregnancy. Females of childbearing potential must be using an effective contraceptive method (e.g., abstinence, prescription oral contraceptives, contraceptive injections, MRI-safe intrauterine device, double-barrier method, male partner sterilization)
* Any contraindications to having an MRI scan, including cardiac pacemakers, metal vascular clips or stents, artificial heart valves, certain kinds of prostheses, brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings (wounded in military combat, sheetmetal workers, welders, and others), transdermal drug delivery systems, and certain tattoos with metallic ink. NOTE: Participants will be screened for these conditions at screening, and will be required to fill out a standard MRI screening form at the Brain Imaging Center, which will be reviewed by an MRI technician prior to each MRI scan
* Scheduled to receive first ECT treatment on a Friday

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twelve study participants between the ages of 18-55 with will be recruited from inpatient units at McLean Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Gln/Glu ratio following the first ECT treatment | Participants will undergo an MR scan within 24 hours of their first ECT treatment
  The Gln/Glu ratio is examined in the anterior cingulate cortex (ACC) and the parieto-occipital cortex (POC) following the first ECT treatment.

SECONDARY OUTCOMES:
The Gln/Glu ratio following the sixth ECT treatment. | Participants will undergo an MR scan within 24 hours of their sixth ECT treatment, which is approximately two weeks after their first ECT treatment
  The Gln/Glu ratio is examined in both the ACC and POC following the sixth ECT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, M.D., Principal Investigator — Mclean Hospital